CLINICAL TRIAL: NCT06577363
Title: Special Drug Use Surveillance of LIVTENCITY Tablets 200mg (All-Case Investigation)
Brief Title: A Survey of Maribavir Tablets in Participants With Cytomegalovirus Infection
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4013; jRCT2031240302 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cytomegalovirus (CMV)
Keywords: Drug Therapy
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maribavir: Maribavir 400 milligrams (mg), tablets, orally twice a day.
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Maribavir tablets

SUMMARY:
This study is a survey in Japan of Maribavir tablets used to treat participants with Cytomegalovirus (CMV) infection refractory to existing anti-CMV therapy in organ transplantation (including hematopoietic stem cell transplantation).

The main aim of the study is to check if treatment with Maribavir can protect Japanese people against CMV infection, and to check side effect from the study treatment. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

During the study, participants with CMV infection will take Maribavir tablets according to their clinic's standard practice. The study doctors will check for side effects from Maribavir tablets for 27 weeks.

ELIGIBILITY:
Inclusion Criteria:

- All participants with Cytomegalovirus (CMV) infection refractory to existing anti-CMV therapy in organ transplantation (including hematopoietic stem cell transplantation).

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2031-08-30 (Estimated); Study Completion 2031-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least One Adverse Drug Reactions (ADRs) | Up to 27 weeks
  An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. Adverse drug reaction refers (ADR) to AE related to administered drug.

SECONDARY OUTCOMES:
Percentage of Participants With Confirmed CMV viremia Clearance | 27 weeks
  Confirmed CMV viremia clearance will be assessed based on plasma CMV DNA concentration in plasma or CMV positive antigen cell in blood.
Percentage of Participants Who Have a Response to CMV, as Assessed by the Investigator | 27 weeks
  Percentage of participants who have a response to CMV, as assessed by the investigator will be reported.
Percentage of Participants With Resistance to Maribavir Treatment | 27 weeks
  Based on treatment and observation in clinical practice, incidence of CMV resistance to this drug is evaluated.
Percentage of Participants With Graft Rejection | 27 weeks
  Percentage of participants With TEAEs of graft rejection will be reported.
Percentage of Participants With Graft-versus-host Disease (GVHD) | 27 weeks
  Percentage of participants with TEAEs of GVHD will be reported.
Percentage of Participants With All-cause Mortality by the End of the Study | 27 weeks
  Percentage of participants who died during the entire study period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/